CLINICAL TRIAL: NCT04945551
Title: Cellular Adaptations to Training in Patients With Type 2 Diabetes
Acronym: TrainAiD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Flemming Dela, Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Training Adaptations in T2D
Record Dates: First submitted 2021-06-07; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Aerobic exercise; Insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Thirty obese patients with (n=15) and without (n=15) type 2 diabetes will be included in the study. Both groups will undergo a 12-week aerobic exercise training intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes (Experimental): Aerobic exercise training
  Interventions: Behavioral: Aerobic exercise training
- Healthy (Experimental): Aerobic exercise training
  Interventions: Behavioral: Aerobic exercise training

INTERVENTIONS:
Behavioral: Aerobic exercise training — 12 weeks intervention period consisting of aerobic exercise training 3 sessions/week, 45 min/session. All training sessions are supervised. Aerobic training is conducted as ergometer bicycle training at an intensity of 70% of maximal oxygen uptake (x2/wk.) and rowing ergometer exercise at 70% of maximal heart rate (x1/wk.). In week 3, 6 and 9 VO2 max is measured to ensure sufficient adjustment of the workload during the training sessions.

SUMMARY:
Physical training can improve metabolic health in patients with insulin resistance and/or type 2 diabetes (T2D). The cellular and molecular changes underlying the improvements in metabolic health are multi-factorial and only partly understood, but most likely involve adaptation at a multi-organ level that includes improvements in skeletal muscle glucose uptake and adipose tissue insulin sensitivity.

The aim of this project is to study the transcriptional differences in skeletal muscle and adipose tissue at baseline and after a 3-month physical training program in obese patients with and without T2D and to use this information to identify novel therapeutic targets for improvement of glucose disposal and insulin sensitivity in patients with T2D.

Thus, the investigators aim to find answers to the question: What is the mechanism behind the effect of physical activity on insulin sensitivity in type 2 diabetes?

DETAILED DESCRIPTION:
Background and aim

Physical training can improve metabolic health in patients with insulin resistance and/or type 2 diabetes (T2D). The cellular and molecular changes underlying the improvements in metabolic health are multi-factorial and only partly understood, but most likely involve adaptation at a multi-organ level that includes improvements in skeletal muscle glucose uptake and adipose tissue insulin sensitivity.

The literature on the effects of an acute bout of exercise on glucose uptake in skeletal muscle is large, but so far, there is a lack of studies investigating the specific molecular basis for the insulin sensitizing effect of regular physical training.

The aim of this project is to study the transcriptional differences in skeletal muscle and adipose tissue at baseline and after a 3-month physical training program in obese patients with and without T2D and to use this information to identify novel therapeutic targets for improvement of glucose disposal and insulin sensitivity in patients with T2D.

Thus, the investigators aim to find answers to the question: What is the mechanism behind the effect of physical activity on insulin sensitivity in type 2 diabetes?

Methods

Thirty obese patients with (n=15) and without (n=15) type 2 diabetes will be included in the study.

Design: Cohort Study Intervention: 12 weeks intervention period consisting of aerobic exercise training 3 sessions/week, 45 min/session. All training sessions are supervised. Aerobic training is conducted as ergometer bicycle training at an intensity of 70% of maximal oxygen uptake (x2/wk.) and rowing ergometer exercise at 70% of maximal heart rate (x1/wk.). In week 3, 6 and 9 VO2max is measured to ensure sufficient adjustment of the workload during the training sessions.

Experimental methods: Before (1-2 weeks) and after the intervention, the following tests and measurements are performed:

Day A: (Overnight fasting. Duration approx. 3 h)

* Dual energy x-ray absorptiometry (DXA) scan (body composition and body fat)
* Graded exercise test on an ergometer bike (maximal fat oxidation rate)
* Maximal oxygen consumption test (VO2max)
* Handgrip strength (by dynamometer)
* Leg power (Power Rig and sit-to-stand test)

Day B: (Overnight fasting. Duration approx. 9 h)

* 2-step euglycemic, hyperinsulinemic clamp
* Muscle biopsy vastus lateralis
* Fat biopsy subcutaneous lower abdomen
* Flow measurements (Femoral artery by Doppler ultrasound and forearm by strain-gauge plethysmography)
* Energy expenditure (ventilated hood method)

Day A and B are repeated after the training intervention has finished.

Analytical methods:

1. Muscle and fat biopsies: Mitochondrial respiratory capacity and reactive oxygen species production. Single nuclei RNA sequencing (snSeq). Fiber type determination and capillarization.
2. Blood samples: Hormones, metabolites and substrates (e.g. insulin, catecholamines, cortisol, glucose, lactate, pyruvate, ketone bodies, cytokines, and myokines). Plasma proteomic/peptidomic analysis.

In summary, this study will reveal cell types and genes in skeletal muscle and adipose tissue that are affected by training and/or that shows differential regulation in patients with T2D versus control subjects.

Statistical considerations:

A power calculation indicates that a significant difference in training induced insulin sensitivity will be detectable when n ≥ 10, based on power = 0.95 and level of significance set to P<0.05. This allows for a dropout rate of a 15-20% with some margin. Mixed model analysis will be used for data analysis of phenotypical data, and bioinformatical tools for the snSeq data and for the interaction between gene- and phenotype expression.

Ethical considerations:

The project was approved by The Regional Ethical Committee of the Capital Region (H-20046605) the 15th of December 2020.

ELIGIBILITY:
Inclusion Criteria:

* Overweight to obese (BMI 28-35 kg/m2)
* Normal resting ECG

Specific for patients with T2D:

* In antiglycemic treatment with diet +/- metformin, SLGT-2 inhibitors, sulfonylurea, GLP1-RA, or DPPV-4 inhibitors
* Time since diagnosis max 4 yrs

Exclusion Criteria:

* Diagnosed with cardiovascular disease (minor to moderate hypertension allowed, defined as prescribed maximally two different antihypertensive drugs)
* Epilepsy
* Kidney disease (GFR<50 ml/min)
* Regular exercise activity
* Inability to perform bicycling and rowing ergometer exercise
* Inability to understand Danish language (written and spoken)

Specific for patients with T2D:

- Insulin treatment

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | Change from baseline at 12 weeks
  Euglycemic hyperinsulinemic clamp
Blood flow | Change from baseline at 12 weeks
  Pulsed-wave Doppler ultrasound (A. femoralis) and venous occlusion strain-gauge plethysmography (forearm)
Gene expression will be quantitatively determined at cellular resolution using single nuclei sequencing | Change from baseline at 12 weeks
  The snSeq data will be analysed using state of the art computational approaches to detect changes in cell type composition and differences in gene expression patterns of specific cell types. These approaches will include: I) normalizations of raw counts; II) feature selection based on most variable genes; III) Conos or Canonical correlation analysis to align the cells across samples; IV) Visualization using dimensionality reduction approaches such as Uniform Approximation and Projection (UMAP) and t-distributed Stochastic Neighbour Embedding (t-SNE); V) RNA velocity and trajectory inference methods to follow changes in cell type identities.

SECONDARY OUTCOMES:
Glucose homeostasis | Change from baseline at 12 weeks
  Changes in HbA1c concentration
Cardiorespiratory fitness | Baseline and after 3, 6, 9 and 12 weeks of aerobic exercise training
  Changes in maximal oxygen uptake

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Dela, MD, DMSc, Principal Investigator — University of Copenhagen
Locations (1):
- Xlab, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Can be provided upon reasonable request